CLINICAL TRIAL: NCT01064349
Title: Breast Cancer With Over-expression of erbB2 Study of the Treatment Paradigm in Metastasis to BRAIN (BRAINSTORM)
Brief Title: Breast Cancer With Over-expression of erbB2-BRAINSTORM
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113349
Record Dates: First submitted 2010-01-21; First posted 2010-02-08 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-05

CONDITIONS: Cancer
Keywords: ErbB2+ breast cancer; ErbB2 treatment; brain metastases
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients with brain metastases: Female Erb2+ breast cancer patients with brain metastases diagnosed between January 2006 and December 2008 in 6 Asian countries (Indonesia, Korea, Malaysia, Philippines, Singapore, and Thailand).
  Interventions: Drug: Anti-erbB2 therapy as part of a treatment regimen for either brain metastases or primary breast cancer

INTERVENTIONS:
Drug: Anti-erbB2 therapy as part of a treatment regimen for either brain metastases or primary breast cancer — Trastuzumab or Lapatinib

SUMMARY:
This retrospective cohort study aims to improve our understanding of the current paradigm for treatment of brain metastases in erbB2+ breast cancer patients in the Asia Pacific region. We aim to identify approximately 300 erbB2+ breast cancer patients with brain metastases diagnosed between 2006-2008 in 6 countries. Medical records will be analyzed to determine the treatment pattern for brain metastases, including anti-erbB2 therapy. Additional objectives are to understand the impact of anti-erbB2 therapy on survival after brain metastases and to investigate the relationship between anti-erbB2 therapy for brain metastases and: 1) the time interval between diagnosis of erb2+ breast cancer and brain metastasis, and 2) the occurrence of brain metastasis as the first site of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with erbB2+ breast cancer. ErbB2 positivity will be as determined by respective institutional standards, and will be based on medical history only.
2. Brain metastasis diagnosis made between January 2006 - December 2008.

Exclusion Criteria:

1. Women who have another primary cancer diagnosed between the time of breast cancer diagnosis and brain metastasis..
2. Patient has leptomeningeal metastases only without parenchymal brain involvement (since this pattern of the disease requires a different treatment approach.)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study aims to enrol approximately 300 Erb2+ breast cancer cases with brain metastases in 6 Asian countries (Indonesia, Korea, Malaysia, Philippines, Singapore, and Thailand).
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2009-05-06; Primary Completion 2011-06-03 (Actual); Study Completion 2011-06-03 (Actual)

PRIMARY OUTCOMES:
To describe the treatment pattern of brain metastasis in ErbB2 over-expressing breast cancer in Asia Pacific countries. | Time (in months) from date of first diagnosis of brain metastasis through to death or end of study period

SECONDARY OUTCOMES:
To describe the survival of ErbB2 over-expressing breast cancer patients with brain metastasis after diagnosis of brain metastasis in relation to the receipt of anti-erbB2 therapy. | Time (in months) from date of first diagnosis of brain metastasis through to death or end of study period
Describe association between usage of anti-erbB2 therapy (before brain metastasis) & 1) time interval from diagnosis of erbB2+ breast cancer to occurrence of brain metastasis and 2) occurrence of brain metastasis as the first site of disease progression | Time (in month) between the date of diagnosis of erbB2+ breast cancer and date of first diagnosis of brain metastasis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Philippines (2):
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Quezon City
- GSK Investigational Site, Singapore, Singapore
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

REFERENCES:
- [Background] Yap YS, Cornelio GH, Devi BC, Khorprasert C, Kim SB, Kim TY, Lee SC, Park YH, Sohn JH, Sutandyo N, Wong DW, Kobayashi M, Landis SH, Yeoh EM, Moon H, Ro J. Brain metastases in Asian HER2-positive breast cancer patients: anti-HER2 treatments and their impact on survival. Br J Cancer. 2012 Sep 25;107(7):1075-82. doi: 10.1038/bjc.2012.346. Epub 2012 Aug 23. PMID 22918394